CLINICAL TRIAL: NCT05838378
Title: The Impact of Cigarillo Warnings on Purchasing and Smoking Behaviors Among Young Adult Cigarillo Users, Aim 2 Survey
Brief Title: Cigarillo Warnings Image Sorting Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Wake Forest University Health Sciences (Other); Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-43316; R01CA260460 (NIH)
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Smoking, Cigar
Keywords: Current cigarillo user; Cigar/cigarillo quit intentions; Pictorial warning format; Surgeon General text warning format; FDA text warning format
MeSH Terms: conditions — Cigar Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pictorial warnings (Experimental): Participants randomized to this group will view pictorial cigarillo warnings.
  Interventions: Other: Package image sorting with pictorial warnings
- FDA text-only warnings (Active Comparator): Participants randomized to this group will view FDA text-only warnings.
  Interventions: Other: Package image sorting with FDA text-only warnings
- Surgeon General text-only warnings (Active Comparator): Participants randomized to this group will view Surgeon General text-only warnings.
  Interventions: Other: Package image sorting with Surgeon General text-only warnings

INTERVENTIONS:
Other: Package image sorting with pictorial warnings — Weekly for four weeks participants will complete an image-sorting task based on sorting cigarillos by flavor categories [fruit (e.g., Grape), alcohol (e.g., Wine) desserts/candy (e.g., Sticky Sweets), mint (e.g., Menthol), color (e.g., Blue Crush), and other]. Participants will sort 18 images of cigarillo packages from various brands with pictorial warnings on each pack.
  Arms: Pictorial warnings
Other: Package image sorting with Surgeon General text-only warnings — Weekly for four weeks participants will complete an image-sorting task based on sorting cigarillos by flavor categories [fruit (e.g., Grape), alcohol (e.g., Wine) desserts/candy (e.g., Sticky Sweets), mint (e.g., Menthol), color (e.g., Blue Crush), and other]. Participants will sort 18 images of cigarillo packages from various brands with Surgeon General text-only warnings on each pack.
  Arms: Surgeon General text-only warnings
Other: Package image sorting with FDA text-only warnings — Weekly for four weeks participants will complete an image-sorting task based on sorting cigarillos by flavor categories [fruit (e.g., Grape), alcohol (e.g., Wine) desserts/candy (e.g., Sticky Sweets), mint (e.g., Menthol), color (e.g., Blue Crush), and other]. Participants will sort 18 images of cigarillo packages from various brands with FDA text-only warnings on each pack.
  Arms: FDA text-only warnings

SUMMARY:
The goal of this study is to examine the impact of repeated exposure to cigarillo warnings on cigarillo users' intentions and behaviors for cigarillo smoking. Eligible participants will be randomized to one of three experimental conditions that will vary based on cigarillo warning format.

For 4 weeks, participants will participate in an image-sorting task where they will be asked to sort a set of ~18 cigarillo packages into flavor categories determined a priori by the research team (e.g., Mint, Fruit, Dessert).

At the end of the study, participants will be notified of the purpose of the study and provided links to resources with information about the harms of cigarillo smoking and cessation.

The study will be conducted in an online survey, working with Qualtrics research company, who will program the survey, recruit and screen participants, and administer the survey.

ELIGIBILITY:
Inclusion Criteria:

* Current cigarillo user-used cigarillos at least one time per week in the past month
* Recruited through Qualtrics Research Services

Exclusion Criteria:

* Not recruited through Qualtrics Research Services
* Non-English speaking

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 764 (Actual)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Intention to quit smoking cigarillos in the next 30 days at baseline | Baseline
  Assessed by the score for 4 survey items: how interested participants are in quitting cigarillo smoking in the next 30 days; how likely they are to quit smoking cigarillos in the next 30 days; how much they plan to quit smoking cigarillos in the next 30 days; and how successful they think they would be if they tried to quit smoking cigarillos in the next 30 days. Each survey item has a 5-pt response scale (1=Not at all to 5= Extremely).Three of the four items will be averaged. Higher scores are associated with a greater intention to quit.
Intention to quit smoking cigarillos in the next 30 days at weeks 2-4 | Weeks 2-4
  Assessed by the score for 4 survey items: how interested participants are in quitting cigarillo smoking in the next 30 days; how likely they are to quit smoking cigarillos in the next 30 days; how much they plan to quit smoking cigarillos in the next 30 days; and how successful they think they would be if they tried to quit smoking cigarillos in the next 30 days. Each survey item has a 5-pt response scale (1=Not at all to 5= Extremely).Three of the four items will be averaged. Higher scores are associated with a greater intention to quit.

SECONDARY OUTCOMES:
Cigarillo smoking behavior in the past week | Baseline, Weeks 2-4
  Assessed by 4 survey items with response options of yes/no: in the past week, have you: 1) butted out a cigarillo before you finished because you wanted to smoke less? 2) stopped yourself from smoking a cigarillo because you wanted to smoke less? 3) tried to quit cigarillos completely; 4) tried cutting back on your cigarillo smoking?

OTHER OUTCOMES:
Quitting self-efficacy based on anticipated success | Baseline, Weeks 2-4
  Assessed by a single survey item asking how successful participants think they would be if they tried to quit smoking in the next 30 days. The survey item has a 5-pt response scale (0=Not at all to 5= Extremely).
Quitting stages of change on a quit ladder | Baseline, Weeks 2-4
  Assessed by an image of a quit ladder, asking participants where they are now on the ladder in regards to cigarillo smoking (1 no thought of quitting - 10 taking action to quit).
Warning recall | Baseline, Weeks 2-4
  Assessed by one survey item asking participants if they noticed any health warnings on the cigarillo packages during the study, with response options of Yes, No, and I'm not sure. Recall is defined as a "Yes" response.
Warning recognition | Baseline, Weeks 2-4
  Assessed by one survey item asking participants to identify which warning they saw during the study period. Participants will be shown their warning, a warning they did not see, and "I don't know" response options. Selecting the correct warning indicates warning recognition.
Warning reactions | Baseline, Weeks 2-4
  Assessed by four survey items assessing participants' perceptions of the warning for 1) grabbing attention; 2) eliciting disgust/emotions; 3) thinking about the risks; 4) self-reported learning. Response options from 1 = not at all to 5 = very much.
Beliefs about harms associated with cigarillo smoking | Baseline, Weeks 2-4
  Assessed by 11 survey items on participant's beliefs about the harms associated with cigarillo smoking, such as relative risk to cigarettes, getting cancer, and inhaling harmful chemicals. 5 point response scale (1=strongly disagree to 5=strongly agree). Higher scores are associated with stronger beliefs about the harms associated with cigarillo smoking.
Knowledge about harms associated with cigarillo smoking | Baseline, Weeks 2-4
  Assessed by 10 survey items on participant's knowledge about the harms associated with cigarillo smoking, such as cigarillos being addictive and causing heart disease with three response options: True, False, I don't know.
Social interactions | Week 4
  Assessed with 3 survey items about: 1) the frequency in which participants talked to others about the harms of cigarillo smoking, 20 quitting cigarillo smoking, or 3) about the packages in the study. Response options range from 1 = never to 5 = 10 times or more.
Warning Relevance | Week 4
  Assessed with 2 survey items about participants' perceptions about the relevance of the cigarillo warning for those who smoke cigarillos with cannabis (i.e., blunts). 5 response options from 1 = not at all to 5 = very much.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ross, PhD, Principal Investigator — School of Public Health - Health Law Policy & Management Dept
Locations (1):
- Boston University School of Public Health, study online, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No